CLINICAL TRIAL: NCT06714019
Title: WI241665 2018 GLOBAL ASPIRE TTR Amyloidosis _ Transthyretin Amyloidosis National Registry - a Prospective Non-interventional, Longitudinal, Observational Multicentre Study
Brief Title: PL_GNT01_ISR_Grant 53234273
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Monika Gawor-Prokopczyk, PhD, National Institute of Cardiology, Warsaw, Poland
Other Study IDs: 53234273
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-05

CONDITIONS: Transthyretin Cardiomyopathy (TTR-CM); Transthyretin (TTR) Amyloid Cardiomyopathy; Transthyretin Amyloidosis
Keywords: transthyretin; transthyretin amyloidosis; ATTR; Transthyretin amyloid cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
We carry out a prospective non-interventional, longitudinal, observational multicentre registry designed to improve our understanding of the epidemiology of TTR amyloidosis in our country. The main objective of the proposed study is to determine the occurrence of TTR amyloidosis and describe clinical profile of patients in the population of our country.

DETAILED DESCRIPTION:
Demographic information, TTR genotype, medical history, family history of the disease, and transplant history are assessed at baseline. On return visits, signs and symptoms of the disease are evaluated, general examinations are conducted, and laboratory data, measures of neurologic and cardiovascular function, and quality of life are assessed according to the standard of care for patients.

Specific Aims and Hypotheses

Our working hypotheses are:

1. TTR amyloidosis affects patients in the population of our country;
2. there are specific TTR mutations in the population of our country;
3. there is genotype-phenotype relationship in hereditary TTR amyloidosis;
4. there are risk factors for TTR amyloidosis in the population of our country. These hypotheses will be tested in our specific aims. In aim 1. we will describe the occurrence of TTR amyloidosis in the population of our country, including the hereditary and acquired forms of the disease.

In aim 2. we will determine and characterize high frequency TTR mutations in the population of our country.

In aim 3. we will determine a clinical profile of patients and we will try to enhance understanding of the natural history of TTR amyloidosis, including the variability, progression of the disease, and predisposing factors. We will evaluate patients' quality of life.

In aim 4. we will search for genotype-phenotype relationship in hereditary TTR amyloidosis.

In aim 5. we will evaluate effects of liver transplantation and other treatments on disease progression in our patients. We will advance knowledge of the disease to optimize the assessment, treatment and monitoring of patients.

In aim 6. we will formulate novel hypotheses for further prospective studies. We will form a community of medical experts on amyloidosis (cardiologists, neurologist, internal medicine physicians, as well as other specialists) to create in the future national centre of amyloidosis in our country that would offer the highest standard of care and gather clinical data on this rare disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old with confirmed diagnosis of TTR amyloidosis

Exclusion Criteria:

* Refusal to participate in the study. Light-chain amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals with wild-type TTR amyloidosis and patients with a confirmed TTR mutation with or without a diagnosis of TTR amyloidosis will be eligible to be enrolled in the registry. Enrolment is voluntary and dependent on each subject's written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
disease progression | From enrollment for at least 12 month
  Signs and symptoms of the disease are evaluated, general examinations are conducted, and laboratory data, measures of neurologic and cardiovascular function, and quality of life are assessed according to the standard of care for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No